CLINICAL TRIAL: NCT04083781
Title: Efficacy and Safety of Concizumab Prophylaxis in Patients With Haemophilia A or B With Inhibitors
Brief Title: Research Study to Look at How Well the Drug Concizumab Works in Your Body if You Have Haemophilia With Inhibitors
Acronym: explorer7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7415-4311; U1111-1225-9670 (Other: World Health Organization (WHO)); 2018-004889-34 (Registry Identifier: European Medicines Agency (EudraCT))
Expanded Access: NCT04921956 (Available)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — concizumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to concizumab prophylaxis (ppx) or no ppx or assigned into non-randomised treatment arms, based on their treatment regimen before entering the trial. Main part of trial is completed when participant has completed at least 24 weeks of participation in arm 1 or 32 weeks in arms 2, 3 and 4. After main part, all participants will be offered to continue in extension part and receive treatment until concizumab is commercially available in their countries or until 31 December 2026 for up to 332 weeks (arms 1-4) or up to 324 weeks (randomised to arm 1 before the pause). After extension part, participant will enter safety follow-up part on visit 26a, which defines end-of-treatment. Participant will receive last dose of trial drug at home on day prior to visit 26a. On visit 26a, participants will either start up commercially available concizumab or revert to previous ppx schedule or on-demand regimen. Follow-up part will start on visit 26a and lasts for 7 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: No prophylaxis (Experimental): Haemophilia A with inhibitors (HAwI) and haemophilia B with inhibitors (HBwI) patients, previously treated on-demand, will be randomised 1:2 to no prophylaxis versus concizumab prophylaxis. In the extension part, patients in arm 1 will receive daily concizumab subcutaneous (s.c., under the skin) injections.
  Interventions: Drug: Concizumab
- Arm 2: Concizumab prophylaxis (Experimental): HAwI and HBwI patients, previously treated on-demand, will be randomised 1:2 to no prophylaxis versus concizumab prophylaxis.
  Interventions: Drug: Concizumab
- Arm 3: Concizumab prophylaxis (Experimental): The HAwI and HBwI patients enrolled into the concizumab phase 2 trial (NN7415-4310) at time of transfer will be offered enrolment into this trial. It is required that these patients are on concizumab prophylaxis up until enrolment into the trial. These patients will continue concizumab prophylaxis.
  Interventions: Drug: Concizumab
- Arm 4: Concizumab prophylaxis (Experimental): Patients previously on prophylaxis with by-passing agents and on-demand patients who are screened at a timepoint where the required number of patients in arms 1 and 2 have been randomised. These patients will, if eligible, be enrolled into the trial and will initiate concizumab prophylaxis at visit 2a (week 0).
  Interventions: Drug: Concizumab

INTERVENTIONS:
Drug: Concizumab — Concizumab will be administered daily subcutaneously (s.c., under the skin). When patients are randomised to concizumab prophylaxis they will receive a loading dose of 1.0 mg/kg concizumab at visit 2a (week 0: arm 2, 3 & 4) or visit 9a (week 24: arm 1) followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week dose adjustment period on 0.20 mg/kg concizumab, the patients can be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab. A potential dose adjustment will take place at visit 4a.1 (week 6: arm 2, 3 & 4) or 9a.3 (week 30: arm 1) and will be based on the concizumab exposure level measured at the previous visit 4a (week 4) or 9a.2 (week 28). Patients who have concizumab exposure levels of 200-4000 ng/mL will stay at 0.20 mg/kg concizumab. Patients in arm 1 will continue on-demand treatment with their usual bypassing product until visit 9a (week 24: end of main part for arm 1).

SUMMARY:
This study will test how well a new medicine called concizumab works in the body of people with haemophilia A or B with inhibitors. The purpose is to show that concizumab can prevent bleeds in the body and is safe to use. Participants who usually only take medicine to treat bleeds (on-demand) will be placed in one of two groups. In one group, participants will get study medicine from the start of the study. In the other group, participants will continue with their normal medicine and get study medicine after 6 months. Which treatment the participant gets is decided by chance. Participants who usually take medicine to prevent bleeds (prophylaxis treatment) or who are already being treated with concizumab (study medicine) will receive the study medicine from the start of the study. Participants will get 1 injection with the study medicine every day under the skin. This participants will have to do themselves and can be done at home. The study doctor will hand out the medicine in the form of a pen-injector. The pen-injector will contain the study medicine. The study will last for about seven years. The length of time the participants will be in the study depends on when they agreed to take part or when the medicine is available for purchase in their country (31 December 2026 at the latest). The time between visits will be approximately 4 weeks for the first 6 to 12 months, depending on the group participants are in and approximately 8 weeks for the rest of the study. Participants will be asked to record information into an electronic diary during the study and may also be asked to wear an activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male aged 12 years or older at the time of signing informed consent.
* Congenital Haemophilia A or B of any severity with documented history of inhibitor (equal to or above 0.6 Bethesda Units (BU).
* Patient has been prescribed, or in need of, treatment with bypassing agents in the last 24 weeks prior to screening (for patients not previously enrolled in NN7415-4310 (explorer 4)).

Exclusion Criteria:

* Known or suspected hypersensitivity to any constituent of the trial product or related products.
* Known inherited or acquired coagulation disorder other than congenital haemophilia.
* Ongoing or planned Immune Tolerance Induction treatment.
* History of thromboembolic disease (includes arterial and venous thrombosis including myocardial infarction, pulmonary embolism, cerebral infarction/thrombosis, deep vein thrombosis, other clinically significant thromboembolic events and peripheral artery occlusion). Current clinical signs of, or treatment for thromboembolic disease. Patients who in the judgement of the investigator are considered at high risk of thromboembolic events (thromboembolic risk factors could include, but are not limited to, hypercholesterolemia, diabetes mellitus, hypertension, obesity, smoking, family history of thromboembolic events, arteriosclerosis, other conditions associated with increased risk of thromboembolic events.)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2027-02-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (95):
- United States (7):
  - Center for Inherited Blood Dis, Orange, California
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - Washington University School of Medicine_St. Louis, St Louis, Missouri
  - St. Jude Affiliate Clinic at Novant Health Hemby Children's, Charlotte, North Carolina
  - TriStar Medical Group Children's Specialist, Nashville, Tennessee
  - University of Texas San Antonio, San Antonio, Texas
- Algeria (2):
  - Haematology and Blood Bank Department, Algiers
  - CHU Constantine BEN BADIS/ Hematology department, Constantine
- Australia (3):
  - The Alfred, Melbourne, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Fiona Stanley Hospital - Haemophilia and Haemostasis Centre, Murdoch, Western Australia
- Klin. Abt. f. Hämatologie und Hämostaseologie, AKH Wien, Vienna, Austria
- UMHAT Tsaritsa Yoanna - ISUL EAD, Pediatric clinical hematology and oncology, Sofia, Bulgaria
- Hamltn Hth Sci/McMstr Child Hosp, Hamilton, Ontario, Canada
- Croatia (2):
  - KBC Zagreb, Rebro, Hemofilija centar, Zagreb
  - KBC Zagreb, Zavod za pedijatrijsku hematologiju, Zagreb
- Czechia (2):
  - Ustav Hematologie a krevni tranfuze, Prague
  - Fakultni nemocnice v Motole, Prague
- Skejby Blodsygdomme, blødercentret, Aarhus N, Denmark
- France (4):
  - Hospices Civils de Lyon- Hopital Louis Pradel, Bron
  - Centre Hospitalier de Clermont-Ferrand-Hopital Estaing, Clermont-Ferrand
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
- India (6):
  - St. John's Medical college and Hospital, Bangalore, Karnataka
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - All India Institute of Medical Sciences_New Dehli, New Dehli, New Delhi
  - CMCV, Ranipet, Tamil Nadu
  - All India Institute of Medical Sciences_New Dehli, New Delhi
- Italy (7):
  - Dipartimento di Ematologia Univ. Firenze, Florence, FI
  - Istituto Oncologico Veneto - Oncoematologia IOV, Castelfranco Veneto
  - Oncoematologia IOV, Castelfranco Veneto
  - Istituto di Medicina Int. A. Bianchi Bonomi Univ. Milano, Milan
  - Azienda OU "S.Maria della Misericordia", Udine
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Donna Bambino Borgo Trento - U.O.C. Oncoematologia Pediatrica, Verona
  - Ospedale Donna Bambino U.O.C. Oncoematologia Pediatrica, Verona
- Japan (7):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Kagoshima City Hospital, Kagoshima
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Mie University Hospital, Mie
  - Nara Medical University Hospital_Pediatrics, Nara
  - Saitama Medical Univ. Hospital, Saitama
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- Malaysia (3):
  - Hospital Pulau Pinang_Georgetown, Penang, George Town, Pulau Pinang
  - Hospital Queen Elizabeth 1, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico
- Rikshospitalet - avdeling for blodsykdommer, Oslo, Norway
- Poland (6):
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki, Oddzial Kliniczny Hematologii, Krakow, Lesser Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - SPSK nr 1 Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
  - Uniwersytecki Szpital Kliniczny nr 1 Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
  - Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego We Wroclawiu, Wroclaw
- ULS São João, E.P.E., Porto, Portugal
- Russia (5):
  - Children Regional Clinical Hospital, Krasnodar
  - Morozovskaya municipal children hospital, Moscow
  - National Medical Research institution of haemotology, Moscow
  - Republican Hospital n.a. V. A. Baranov, Petrozavodsk
  - City out-patient clinic 37, City Hemophilia Centre, Saint Petersburg
- Serbia (5):
  - Clinical Centre of Serbia, Institute for Haematology, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
  - University Clinical Centre Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
  - Institute for Health Care of Children and Adolescents, Novi Sad
- Nemocnica sv. Cyrila a Metoda, UNB,Klinika hemat. a transfuz, Bratislava, Slovakia
- South Africa (3):
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
  - Haematology Clinic, Durban, KwaZulu-Natal
  - Pietersburg Hospital, Polokwane, Limpopo
- South Korea (2):
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (7):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Univ. Central de Asturias, Oviedo
  - Hospital Virgen del Rocío, Seville
- Sweden (2):
  - Koagulationsmottagning, Malmo
  - Koagulationsmottagningen, Solna
- Thailand (3):
  - Sunpasitthiprasong Hospital_Pediatrics Department, Ubon Ratchathani, Mueang Distirct,
  - Ramathibodi Hospital_Department of Haematology, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital _Pediatric Hematology and Oncology, Chiang Mai
- Turkey (Türkiye) (4):
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Onkoloji Enstitüsü, Capa-ISTANBUL, Capa-ISTANBUL
  - Akdeniz Üniversitesi Hastanesi- Hematoloji, Antalya, Konyaaltı/ Antalya
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Hematoloji, Adana
- Ukraine (2):
  - National specialized children's hospital 'OHMATDYT' - Haemostasis centre, Kyiv
  - Institute of blood pathology and transfusion medicine of NAMSU - General and haematol. surgery, Lviv
- United Kingdom (5):
  - West Midlands Adult Comprehensive Care Haemophilia, Birmingham
  - Great Ormond Street Hospital for Children, London
  - Manchester Royal Infirmary_Manchester, Manchester
  - Queen's Medical Centre - Haemophilia Comprehensive Care Centre, Nottingham
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Mahlangu J, Boban A, Bruzelius M, Castaman G, Hampton KK, Knoebl P, Lebreton A, Linari S, Lopez-Jaime FJ, Tavares CMMT, Nekkal MS, Nogami K, Nielsen ARH, Shapiro AD, D'Oiron R. Concizumab in hemophilia with inhibitors: Longer-term efficacy and safety results from the phase 3 explorer7 study. Blood Adv. 2026 Jan 7:bloodadvances.2025018264. doi: 10.1182/bloodadvances.2025018264. Online ahead of print. PMID 41499759
- [Derived] Tran H, von Mackensen S, Abraham A, Castaman G, Hampton K, Knoebl P, Linari S, Odgaard-Jensen J, Neergaard JS, Stasyshyn O, Thaung Zaw JJ, Zulfikar B, Shapiro A. Concizumab prophylaxis in persons with hemophilia A or B with inhibitors: patient-reported outcome results from the phase 3 explorer7 study. Res Pract Thromb Haemost. 2024 Jun 17;8(4):102476. doi: 10.1016/j.rpth.2024.102476. eCollection 2024 May. PMID 39099801
- [Derived] Matsushita T, Shapiro A, Abraham A, Angchaisuksiri P, Castaman G, Cepo K, d'Oiron R, Frei-Jones M, Goh AS, Haaning J, Hald Jacobsen S, Mahlangu J, Mathias M, Nogami K, Skovgaard Rasmussen J, Stasyshyn O, Tran H, Vilchevska K, Villarreal Martinez L, Windyga J, You CW, Zozulya N, Zulfikar B, Jimenez-Yuste V; explorer7 Investigators. Phase 3 Trial of Concizumab in Hemophilia with Inhibitors. N Engl J Med. 2023 Aug 31;389(9):783-794. doi: 10.1056/NEJMoa2216455. PMID 37646676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 27 countries. There were 70 sites that randomised participants. The details are as follows: Algeria (2), Australia (2), Austria (1), Bulgaria (1), Canada (0), Croatia (1), Czech Republic (1), Denmark (1), France (4), India (4), Italy (4), Japan (6), Republic of Korea (2), Malaysia (3), Mexico (1), Poland (4), Portugal (1), Russian Federation (5), Serbia (1), South Africa (2), Spain (5), Sweden (1), Thailand (3), Turkey (4), Ukraine (2), UK (3), United States (6).
Pre-assignment Details: 133 participants were actually randomised for the study. The data presented in the results form is till the 56 week cut off (except the data for primary outcome measure, patient reported outcome measures, maximum concizumab plasma concentration and area under the concizumab plasma concentration-time curve) as the study is still ongoing with the extension phase.
Groups:
- Arm 1: Previous on Demand: No Prophylaxis: Participants with hemophilia A with inhibitor (HAwI) and hemophilia B with inhibitor (HAwB) received their on-demand treatment for a minimum of 24 weeks. Subsequently, following the main phase, participants transitioned to the new dosing regimen for concizumab and were scheduled to undergo concizumab prophylaxis in the trial's extension phase.
- Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX): Participants with HAwI and HBwI received a loading dose of 1.0 milligrams per kilograms (mg/kg) concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg.
- Arm 3: Concizumab Non-naive: Concizumab PPX: Participants with HAwI and HBwI received a loading dose (participants entering from the phase 2 trial [N7415-4310] were not to receive a loading dose) of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg.
- Arm 4: Concizumab Naive: Concizumab PPX: Participants with HAwI and HBwI received a loading dose of 1.0 mg/kg concizumab subcutaneously followed by an initial daily dose of 0.20 mg/kg concizumab from treatment day 2. Within an initial 5-8-week maintenance dose setting period on 0.20 mg/kg concizumab, the participants could be increased or decreased in dose to 0.25 mg/kg or 0.15 mg/kg concizumab or stayed at 0.20mg/kg.
Period: Main Part
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Started | 19 | 33 | 21 | 60
Full Analysis Set (FAS) | 19 | 33 | 21 | 60
Safety Analysis Set (SAS) | 19 | 33 | 21 | 60
Completed | 13 | 27 | 15 | 53
Not Completed | 6 | 6 | 6 | 7
Not completed — Physician Decision | 0 | 1 | 2 | 0
Not completed — Death | 1 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 3 | 7
Period: Extension Part
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Started | 13 | 27 | 15 | 53
Completed | 0 | 0 | 0 | 0
Not Completed | 13 | 27 | 15 | 53
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Ongoing | 13 | 25 | 15 | 51

BASELINE CHARACTERISTICS:
Population: Baseline characteristic data is reported for on-treatment without data on initial regimen (OTexIR) analysis set which included the time period where participants were considered to be affected by on-demand treatment or treatment with the new concizumab dosing regimen excluding observation time during the initial concizumab PPX regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX | Total
Number analyzed (Participants) | 19 | 29 | 15 | 55 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (17.6) | 24.8 (14.4) | 35.1 (10.0) | 26.4 (11.5) | 28.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 19 | 29 | 15 | 55 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 2 | 6
  Not Hispanic or Latino | 16 | 25 | 15 | 52 | 108
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 3
  Asian | 6 | 13 | 4 | 12 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 3 | 8
  White | 9 | 9 | 11 | 38 | 67
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate of Treated Spontaneous and Traumatic Bleeding Episodes
Description: Rate of treated spontaneous and traumatic bleeding episodes is presented. The observation period used for reporting this endpoint is on-treatment without ancillary therapy excl. data on initial regimen for participants exposed to both regimens (OTwoATexIR). It is defined as the time period where participants are treated by either the new concizumab dosing regimen or the initial concizumab dosing regimen (only included if not exposed to the new concizumab dosing regimen) or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleed during any of the cases. The data is reported in the terms of annualised bleeding rate (ABR). Week 0 is defined as time of randomisation to on-demand administration or time of start of the new concizumab dosing regimen.
Time Frame: On demand (arm 1): From week 0 up until start of concizumab treatment (at least 24 weeks) Concizumab (arm 2): From week 0 up until the primary analysis cut-off (at least 32 weeks)
Population: Full analysis set (FAS) included all participants randomised to concizumab prophylaxis (PPX) or on-demand treatment or allocated to arms 3 or 4. This endpoint is only defined for arms 1 and 2 as per protocol.
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX)
Number analyzed (Participants) | 19 | 33
Events per year | 9.8 [6.5 to 20.2] | 0.0 [0.0 to 3.3]
Statistical Analysis 1: Comparison: Arm 1: Previous on Demand: No Prophylaxis vs Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX); Test type: Superiority — Analyses of count endpoints were analysed using a negative binomial regression model with the logarithm of the length of the observation period included (in years) as an offset with randomised treatment regimen, type of haemophilia (HAwI or HBwI) and bleeding frequency (less than 9 or greater than or equal to 9 bleeding episodes during the past 24 weeks prior to screening) as factors comparing arm 1 (on-demand treatment) and arm 2; p < 0.001, Two-sided test of no difference from 1; Annualised bleeding rate ratio = 0.14, 95% CI 2-sided [0.07 to 0.29]

2. Secondary Outcome: Rate of Treated Spontaneous Bleeding Episodes
Description: Rate of treated spontaneous bleeding episodes is presented. The observation period used for reporting this endpoint is OTwoATexIR. It is defined as the time period where participants are treated by either the new concizumab dosing regimen or the initial concizumab dosing regimen (only included if not exposed to the new concizumab dosing regimen) or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleed during any of the cases. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration or time of start of the new concizumab dosing regimen.
Time Frame: On demand (arm 1): From week 0 up until start of concizumab treatment (at least 24 weeks) Extension concizumab (arm 1): From start of new concizumab dosing regimen (week 25) up until week 56 cut-off Concizumab (arm 2): From week 0 up until week 56 cut-off
Population: FAS included all participants randomised to concizumab prophylaxis (PPX) or on-demand treatment or allocated to arms 3 or 4. This endpoint is only defined for arms 1 and 2 as per protocol.
Measure: Median (Inter-Quartile Range); unit: Events per year
Groups:
- Extension Arm 1: Previous on Demand: No Prophylaxis: Participants who completed at least 24 weeks of on demand treatment started with the new concizumab dosing regimen and were planned to receive concizumab prophylaxis (PPX) in the extension part of the trial.
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX)
Number analyzed (Participants) | 19 | 13 | 33
Events per year | 8.4 [3.9 to 14.3] | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 2.2]

3. Secondary Outcome: Rate of Treated Spontaneous and Traumatic Joint Bleeds
Description: Rate of treated spontaneous and traumatic joint bleeds is presented. Observation period used for reporting this endpoint is OTwoATexIR. It is defined as time period where participants are treated by either the new concizumab dosing regimen or the initial concizumab dosing regimen (only included if not exposed to the new concizumab dosing regimen) or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleed during any of the cases. The data is reported in the terms of ABR. Week 0 is defined as time of randomisation to on-demand administration or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX)
Number analyzed (Participants) | 19 | 13 | 33
Events per year | 6.5 [3.2 to 13.1] | 1.3 [0.0 to 1.6] | 0.7 [0.0 to 2.8]

4. Secondary Outcome: Rate of Treated Spontaneous and Traumatic Target Joint Bleeds
Description: Rate of treated spontaneous and traumatic target joint bleeds is presented. Observation period used for reporting the endpoint is OTwoATexIR. It is defined as time period where participants are treated by either the new concizumab dosing regimen or the initial concizumab dosing regimen (only included if not exposed to new concizumab dosing regimen) or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleed during any of the cases. The data is reported in terms of ABR. Week 0 is defined as time of randomisation to on-demand administration or time of start of the new concizumab dosing regimen.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX)
Number analyzed (Participants) | 19 | 13 | 33
Events per year | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

5. Secondary Outcome: Change in 36-item Short Form Health Survey (SF-36v2) Bodily Pain
Description: Change in 36-item SF-36v2 bodily pain from baseline (week 0) to week 24 is presented. SF-36 v2 Health Survey is 36-item generic patient-reported outcome (PRO) instrument measuring health-related quality of life and general health status across disease areas. SF-36 v2 scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and an SD of 10. Lowest and highest scores for bodily pain are 21.68 to 62.0. Higher values indicate better functional health and well-being. Observation period for reporting the data is on-treatment without data on initial regimen (OTexIR) which is defined as time period where participants are considered affected by on demand treatment or treatment with new concizumab dosing regimen. Week 0 is defined as time of randomisation to on-demand administration or start of new concizumab dosing regimen.
Time Frame: Baseline (week 0), Week 24
Population: FAS included all participants randomised to concizumab prophylaxis (PPX) or on-demand treatment or allocated to arms 3 or 4. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 7 | 21 | 13 | 32
Score on a scale | 3.2 (10.1) | 9.3 (9.2) | 4.3 (10.1) | 6.5 (10.0)

6. Secondary Outcome: Change in SF36v2 Physical Functioning
Description: Change in 36-item SF-36v2 physical functioning from baseline (week 0) to week 24 is presented. SF-36 v2 Health Survey is 36-item generic PRO instrument measuring health-related quality of life and general health status across disease areas. SF-36 v2 scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and an SD of 10. Lowest and highest scores for physical functioning are 19.26 to 57.54. Higher values indicate better functional health and well-being. Observation period used for reporting the data is OTexIR which is defined as time period where participants are considered affected by on demand treatment or treatment with new concizumab dosing regimen. Week 0 is defined as time of randomisation to on-demand administration or start of new concizumab dosing regimen.
Time Frame: Baseline (week 0), Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 7 | 21 | 13 | 32
Score on a scale | 1.6 (10.9) | 3.1 (6.2) | 3.8 (8.7) | 4.9 (6.7)

7. Secondary Outcome: Number of Thromboembolic Events
Description: Number of thromboembolic events is presented. The observation period used for reporting the endpoint is on-treatment period which is defined as the time period where participants are considered to be affected by on-demand treatment or concizumab treatment.
Time Frame: On demand (arm 1 ): From week 0 until start of concizumab treatment (atleast 24 weeks) Concizumab (arms 2-4): From week 0 up until week 56 cut-off Extension Concizumab (arm 1): From start of new concizumab dosing regimen (week 25) up until week 56 cut-off
Population: Safety analysis set (SAS) included all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: Events
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 19 | 13 | 33 | 21 | 60
Events | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Number of Thromboembolic Events
Description: as for outcome 7
Time Frame: From week 0 to end of trial (week 167)
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Number of Hypersensitivity Type Reactions
Description: Number of hypersensitivity type reactions is presented. The observation period used for reporting the endpoint is on-treatment period which is defined as the time period where participants are considered to be affected by on-demand treatment or concizumab treatment.
Time Frame: as for outcome 7
Population: SAS included all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: Reactions
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 19 | 13 | 33 | 21 | 60
Reactions | 0 | 0 | 1 | 0 | 1

10. Secondary Outcome: Number of Hypersensitivity Type Reactions
Description: as for outcome 9
Time Frame: From week 0 to end of trial (week 167)
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Number of Injection Site Reactions
Description: Number of injection site reactions is presented. The observation period used for reporting the endpoint is on-treatment period which is defined as the time period where participants are considered to be affected by on-demand treatment or concizumab treatment.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Number; unit: Reactions
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 19 | 13 | 33 | 21 | 60
Reactions | 0 | 1 | 11 | 5 | 43

12. Secondary Outcome: Number of Injection Site Reactions
Description: as for outcome 11
Time Frame: From week 0 to end of trial (week 167)
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Number of Participants With Antibodies to Concizumab
Description: Number of participants with antibodies to concizumab is presented. The observation period used for reporting the endpoint is on-treatment period which is defined as the time period where participants are considered to be affected by on-demand treatment or concizumab treatment.
Time Frame: Concizumab (arms 2-4): From week 0 up until week 56 cut-off Extension Concizumab (arm 1): From start of new concizumab dosing regimen (week 25) up until week 56 cut-off
Population: SAS included all participants exposed to concizumab PPX or randomised to on-demand treatment. The data is presented in a combined manner across all Concizumab PPX arms (arm 2-4) and extension part of concizumab (arm 1) considering that the trial is still ongoing, and that incidence of immunogenicity can still change when the trial is completed, hence it was decided to provide now only total incidence. A more granular picture of immunogenicity per arm, will be provided once trial is finished.
Measure: Count of Participants; unit: Participants
Groups:
- Concizumab PPX: All the participants from extension concizumab (arm 1) and concizumab PPX (arm 2-4) were collectively analysed for the outcome "Number of participants with antibodies to concizumab"
Arm/Group | Concizumab PPX
Number analyzed (Participants) | 127
Participants | 35

14. Secondary Outcome: Number of Participants With Antibodies to Concizumab
Description: as for outcome 13
Time Frame: From week 0 to end of trial (week 167)
Reporting Status: Not Posted, anticipated posting 2026-12

15. Secondary Outcome: Pre-dose (Trough) Concizumab Plasma Concentration (Ctrough)
Description: Pre-dose (trough) concizumab plasma concentration is presented. The observation period used for reporting the endpoint is OTexIR. It is defined as the time period where participants are considered to be affected by on demand treatment or treatment with the new concizumab dosing regimen.
Time Frame: Pre-dose (prior to concizumab administration at week 56)
Population: SAS included all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analyzed = participants with available data for this outcome measure. The endpoint is applicable for reported arms (extension part arm 1, arm 2, arm 3 and arm 4) only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 9 | 24 | 14 | 49
nanograms per milliliter (ng/mL) | 808.7 (263.4) | 570.9 (225.7) | 590.6 (600.9) | 717.3 (328.5)

16. Secondary Outcome: Pre-dose Thrombin Peak
Description: Pre-dose thrombin peak for concizumab is presented. The observation period used for reporting the endpoint is OTexIR. It is defined as the time period where participants are considered to be affected by on demand treatment or treatment with the new concizumab dosing regimen.
Time Frame: Pre-dose (prior to concizumab administration at week 56)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 3 | 11 | 12 | 13
nanomoles per liter (nmol/L) | 104.2 (39.0) | 67.3 (88.7) | 76.2 (78.6) | 75.3 (43.1)

17. Secondary Outcome: Pre-dose Free Tissue Factor Pathway Inhibitor (TFPI) Concentration
Description: Pre-dose free TFPI concentration for concizumab is presented. The observation period used for reporting the endpoint is OTexIR. It is defined as the time period where participants are considered to be affected by on demand treatment or treatment with the new concizumab dosing regimen.
Time Frame: Pre-dose (prior to concizumab administration at week 56)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 9 | 24 | 14 | 49
ng/mL | 13.2 (106.4) | 15.2 (108.7) | 12.1 (123.0) | 11.0 (95.6)

18. Secondary Outcome: Maximum Concizumab Plasma Concentration (Cmax)
Description: Maximum concizumab plasma concentration is presented. The observation period used for reporting the endpoint is on OTexIR. It is defined as the time period where participants are considered to be affected by on demand treatment or treatment with the new concizumab dosing regimen.
Time Frame: Week 24: Predose, 3 hours (h), 6h, 9h, 24h
Population: SAS included all participants exposed to concizumab PPX or randomised to on-demand treatment. Overall number of participants analyzed = participants with available data for this outcome measure. This endpoint is applicable for reported arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 18 | 13 | 38
ng/mL | 992.2 (1.0) | 1514.1 (1.7) | 1153.0 (1.3)

19. Secondary Outcome: Area Under the Concizumab Plasma Concentration-time Curve (AUC)
Description: Area under the concizumab plasma concentration-time curve is presented. The observation period used for reporting the endpoint is OTexIR. It is defined as the time period where participants are considered to be affected by on demand treatment or treatment with the new concizumab dosing regimen.
Time Frame: Week 24: Predose, 3 hours (h), 6h, 9h, 24h
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
Number analyzed (Participants) | 18 | 13 | 38
nanogram*hour per milliliter (ng*hr/mL) | 25991.5 (17069.7) | 47149.3 (38192.8) | 32903.5 (32741.2)

ADVERSE EVENTS:
Time Frame: Up to week 56 cut-off
Description: Safety analysis set (SAS) included all participants exposed to concizumab prophylaxis (PPX) or randomised to no PPX. All presented AEs were treatment emergent AEs (TEAEs). TEAEs were defined as AEs which initiated or worsened during the time period where participants were considered to be affected by on demand treatment or concizumab treatment.
Arm/Group | Arm 1: Previous on Demand: No Prophylaxis | Extension Arm 1: Previous on Demand: No Prophylaxis | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) | Arm 3: Concizumab Non-naive: Concizumab PPX | Arm 4: Concizumab Naive: Concizumab PPX
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/13 | 4/33 | 1/21 | 1/60
Serious Adverse Events (participants affected / at risk) | 3/19 | 2/13 | 9/33 | 2/21 | 9/60
Other Adverse Events (participants affected / at risk) | 8/19 | 8/13 | 15/33 | 13/21 | 35/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Previous on Demand: No Prophylaxis (N=19) | Extension Arm 1: Previous on Demand: No Prophylaxis (N=13) | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) (N=33) | Arm 3: Concizumab Non-naive: Concizumab PPX (N=21) | Arm 4: Concizumab Naive: Concizumab PPX (N=60)
Alcoholic coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin fragment 1.2 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Previous on Demand: No Prophylaxis (N=19) | Extension Arm 1: Previous on Demand: No Prophylaxis (N=13) | Arm 2: Previous on Demand: Concizumab Prophylaxis (PPX) (N=33) | Arm 3: Concizumab Non-naive: Concizumab PPX (N=21) | Arm 4: Concizumab Naive: Concizumab PPX (N=60)
Acarodermatitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (10) | 10 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (2) | 2 (3) | 5 (5) | 5 (5)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (10)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (9)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (11)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Prothrombin fragment 1.2 increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 4 (5)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a pause in the concizumab clinical development programme during the period from March to August 2020, while thromboembolic events were investigated. As of 19 March 2020, all participants on concizumab had stopped treatment and switched to another available treatment as per investigator's discretion. Based on the investigation, risk mitigation actions (including new concizumab dosing regimen) were implemented and trial protocols updated before resuming.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04083781/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT04083781/SAP_001.pdf